CLINICAL TRIAL: NCT03702348
Title: Effect of a Resistance Exercise Program on the Functionality of Individuals With Chikungunya Fever: Randomized Clinical Trial
Brief Title: Resistance Exercise Program on the Functionality of Individuals With Chikungunya Fever
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Isabel Lins Neumann, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1216-9761
Record Dates: First submitted 2018-07-09; First posted 2018-10-11 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Chikungunya Fever
MeSH Terms: conditions — Chikungunya Fever | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise group (Experimental): Progressive resistance exercise protocol with elastic resistance to strengthen the muscle groups that stabilize the main joints affected by Chikungunya Fever. The sessions will be 2 times a week for 12 weeks.
  Interventions: Other: Resistance exercise
- Control group (No Intervention): No intervention during the 12 weeks, being contacted through telephone calls. After the reevaluation at the end of the 12 weeks, this group will perform the same protocol as the experimental group

INTERVENTIONS:
Other: Resistance exercise — Protocol with 5min warm-up exercise and 8 exercises that progress in positioning and resistance based on maximum repetition test. The exercises strengthen both the lower and upper limbs and are intended to simulate activities such as sitting and standing up, climbing stairs, picking up weight ...
  Other Names: Resistance exercise protocol
  Arms: Resistance exercise group

SUMMARY:
Common symptoms of chikungunya fever are persistent arthritis and arthralgia, such symptoms can lead to impairment in functionality. The objective of this study is to evaluate the efficacy of a resistance exercise protocol on the functionality of individuals with chronic musculoskeletal manifestations of Chikungunya fever. Quality of life, number of painful joints, intensity of pain, number of recurrence of exacerbation and thermography are secondary outcomes that will also be evaluated. The protocol uses elastic resistance to strengthen muscle groups that stabilize the main joints affected by Chikungunya Fever. The sessions will be 2 times a week for 12 weeks. The control group will not be submitted to the intervention during the 12 weeks, being contacted through telephone calls. After the reevaluation at the end of the 12 weeks the control group will perform the same protocol. The sample will be characterized and the effect size and the mean difference will be calculated. Intention-to-treat analysis and rate of adherence will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chikungunya fever for more than three months
* Present musculoskeletal symptoms after infection (eg, arthritis or arthralgia)

Exclusion Criteria:

* Cognitive deficit that compromises the understanding and accomplishment of the protocol (MiniMental<24);
* Self-reported disease that contraindicates the performance of research procedures (eg, unstable angina);
* Self-reported diagnosis of neurological disease;
* Prior self-reported diagnosis of other inflammatory or autoimmune rheumatic diseases or fibromyalgia;
* Pregnancy;
* Physical impairment that prevents arrival to the research site or execution of the exercises (eg, use of walking devices);
* Execution of other physiotherapeutic treatments during the research period;
* Regular practice of physical exercises in other places during the period of participation in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in functionality through a walk test | Assessed before intervention, in 6 weeks and after the 12-week intervention
  Performance in seconds of the 40m Fast-paced Walk Test, the longer the time in seconds, the worse the outcome. The normative values for women between 50´s and 60´s age range are 19,90 to 22,60 seconds, and for men in the same age range between 19,32 and 20,73 seconds.
Change in functionality through a stair climb test | Assessed before intervention, in 6 weeks and after the 12-week intervention
  Performance in seconds of the 4 step stair climb test, the longer the time in seconds, the worse the outcome. The normative values mean for healthy women is 10.22 seconds and healthy men is 8.72 seconds
Change in functionality through a chair stand test | Assessed before intervention, in 6 weeks and after the 12-week intervention
  Performance in number of time the patient stands in the 30-Second Chair Stand Test, the higher the number of the better the outcome, the mean for women in the 60´s age range is from 11 to 17 times and for men in the same age range is from 12 to 19 times
Change in functionality of upper limbs | Assessed before intervention, in 6 weeks and after the 12-week intervention
  Function of upper limb trough specific score of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire with 30 items with responses range from 1(not limited) to 5 (extremely limited) and two optional sections, responses are used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability)

SECONDARY OUTCOMES:
Change of score on the Medical Outcomes Study 36 - Item Short - Form Health Survey questionnaire | assessed before intervention, in 6 weeks and after the 12-week intervention
  quality of life assesment through Medical Outcomes Study 36 - Item Short - Form Health Survey questionnaire that consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0 (maximum disability) to 100(no disability) scale
Change in the intensity of pain: VAS | assessed in every intervention day (twice a week for 12 weeks)
  number correspondent to the intensity of pain using visual analogic scale from 0(no pain) to 10 (maximum pain)
Change in the number of painful joints | assessed before intervention, in 6 weeks and after the 12-week intervention
  assessed though a tender joints count, the higher the number the worse the outcome
Change in the number of exacerbation recurrences | assessed through the 12-week intervention period
  the higher the number the worse the outcome
Change in temperature of areas of interest (joints) | assessed before intervention, in 6 weeks and after the 12-week intervention
  assessed with thermography through index of thermic distribution seen through software FLIR Tools 5.3. the higher the temperature the worse the outcome
Change in patients global impression of change | assessed before intervention, in 6 weeks and after the 12-week intervention
  number corresponding to answer of the Patient Global Impression of Change (PGIC) questionnaire being 1 (no change) the worst outcome and 7 (a lot better) the best outcome
Number of patients reporting adverse effects | Reported through study completion, an average of 1 year
  Unexpected effects reported by patients potentially associated with the intervention such as worsening pain, swelling, stiffness or other
Change in muscle strength | Assessed every two weeks during the 12-week intervention period
  Performance in the repetition maximum test (1RM) for every exercise, the higher the value the better the outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Escola de Fisioterapia - UFPE, Recife, Pernambuco, Brazil